CLINICAL TRIAL: NCT03151161
Title: A Prospective,Multi-center, Open-labeled Phase 2 Randomized and Comparative Clinical Study of First Line Intermittent and Maintenance of Icotinib in Combination With Pemetrexed/Carboplatin Compared With Icotinib Single Drug in ⅢB/IV Non Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutation
Brief Title: Intermittent and Maintenance of Icotinib in Combination With Pemetrexed/Carboplatin Compared With Icotinib Single Drug in Ⅲb/IV Non Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201512001
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Lung, Carcinoma
Keywords: chemotherapy; maintenance therapy; icotinib
MeSH Terms: conditions — Lung Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): 1. Chemotherapy regime: Pemetrexed (500mg/m2) + Carboplatin (AUC=5), 1 cycle every 3 weeks, maximum 4 cycles;
  2. Intermittent regime: Icotinib 125mg, three times a day, d2-15 in each cycle; maintenance regime: icotinib 125mg, three times a day, since the last cycle until disease progression.
  Interventions: Drug: Icotinib,Pemetrexed,Carboplatin
- Control Group (Active Comparator): Single drug: Icotinib 125mg, three times a day, continous until disease progression
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib,Pemetrexed,Carboplatin — Pemetrexed (500mg/m2) + Carboplatin (AUC=5), every 3 weeks, maximum 4 cycles; icotinib 125mg, three times a day, d2-15 in each cycle, and icotinib 125mg,three times a day, since the last cycle until disease progression
  Arms: Experimental Group
Drug: Icotinib — Single drug: Icotinib 125mg, three times a day, continuous until disease progression.
  Arms: Control Group

SUMMARY:
EGFR-tyrosine kinase inhibitor(TKI)- ie, erlotinib, gefitinib, icotinib,has been recommended as the first option for EGFR-mutated IIIb/IV NSCLC by serial trials as it prolonged patients' progression-free survival. The OPTIMAl trial indicated that those who received TKI and chemotherapy during the whole treatment window survived longest. Unfortunately, previous studies(INTACT, TRIBUTE et al) that concurrently combined TKI and cytotoxic regimens failed to improve survival in unselected patients. To avoid the potential synergistic antagonism, the FAST-ACT II trial committed a sequential strategy and find a superiority in the combination arm upon chemotherapy even in EGFR-mutated group. However, pharmaceutically, the continuous administration of an EGFR-TKI before subsequent chemotherapy in FAST-ACT II could obviate the effects of cytotoxic agents due to the erlotinib-induced G1 arrest.

On the basis of these and other studies, the investigators hypothesized that a better sequential combination strategy of EGFR-TKI and chemotherapy (adding a EGFR-TKI wash-out window before chemotherapy) would be more efficacious than chemotherapy alone. In this study, the investigators investigate the efficacy(PFS:progression free survival), safety, and adverse-event profile of chemotherapy plus intermittent and maintenance of icotinib compared with icotinib single drug, when these drugs were used as first-line treatment in who had non-squamous lung carcinoma with EGFR gene mutation in China.

ELIGIBILITY:
Inclusion Criteria:

* Present with histologically proven diagnosis of non-Squamous NSCLC Stage IIIB or IV as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer, that is not amenable to curative therapy, such as surgery or radiotherapy and so on.
* Confirmed activating mutation of EGFR-ie, an exon 19 deletion or an exon 21 L858R point mutation.
* Measurable lesions according to RECIST 1.1 criteria.
* Patients between 18 and 75 years of age.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* Estimated life expectancy of ≥12 weeks.
* Haematological stable: ANC > 1.5; PLT > 100; HGB > 90 g/L.
* Adequate liver function: total bilirubin < 1.5 x ULN; AST and ALT < 2.5 x ULN (without liver metastasis); or AST and ALT < 5 x ULN (with liver metastasis).
* Adequate renal function: creatinine < 1.5 x ULN; CCR >= 50ml/min; and urine protein < 2+; for the patients with urine protein >= 2+, 24 hours total urine protein <= 1g.
* INR <= 1.5; aPTT < 1.5 x ULN, within 7 days before treatment.
* For female patients, pregnancy test (blood or urine) needs to be done within 7 days before treatment; if negative, patients need to be consented for proper contraception throughout the treatment and 8 weeks after the completion of treatment. For male patients, they also need to be consented for proper contraception throughout the treatment and 8 weeks after the completion of treatment.
* Signed informed consent document on file.
* Patient compliance and geographic proximity that allow adequate follow up.

Exclusion Criteria:

* Histology is confirmed to be squamous cell carcinoma, mixed NSCLC and SCLC, or squamous cell carcinoma dominant adenosquamous carcinoma.
* Patients previously had targeting HER therapy, including erlotinib, gefitinib, cetuximab，trastuzumab, etc.
* Patients previously had systemic therapy for NSCLC before study, including cytotoxic medicine, target therapy, or other medicines in a clinical trial.
* Physiological incompetence with upper gastrointestinal tract, or malabsorption syndrome, or intolerance of oral drugs, or active peptic ulceration.
* Clinically moderate to severe COPD, active ILD or other pulmonary diseases defined by researchers.
* Uncontrolled ocular inflammation or infection, or other conditions that could lead to ocular inflammation or infection.
* Conditions or risk factors that contraindicate the research medicines.
* Any unsteady systematic diseases, including active infection, uncontrolled high blood pressure, unstable angina, recent angina (within 3 months), congestive heart failure, ischemic heart diseases (within 6 months), severe arrhythmia， severe liver/renal/metabolic diseases.
* Known HIV infection.
* Unhealed wound, active peptic ulceration or fracture.
* Pregnancy or lactation.
* Female patients who refuse contraception throughout treatment and 6 months after the treatment; male patients who refuse contraception throughout treatment and 90 days after the treatment.
* Known severe hypersensitivity to Icotinib, Pemetrexed or Carboplatin.
* Patients with esophago-tracheal fistula.
* Pleural effusion or pericardiac effusion that cannot be controlled by drainage or other procedures.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* Patients had other malignancies apart from NSCLC, except cervical cancer in situ, skin basal cell carcinoma or squamous cell carcinoma, prostate cancer or breast ductal carcinoma in situ that have been adequately treated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 | eight weeks
  Patients were images with computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (1):
- Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided